CLINICAL TRIAL: NCT01442896
Title: STudy to Assess Rapid Disease Progression by Clinical and Genetic Factors In Glaucoma patientS That Are High Risk (STARFISH)
Brief Title: STudy to Assess Rapid Disease Progression by Clinical and Genetic Factors In Glaucoma patientS That Are High Risk
Acronym: STARFISH
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Weinreb, Chairman & Professor of Ophthalmology, University of California, San Diego
Other Study IDs: 111223
Record Dates: First submitted 2011-09-26; First posted 2011-09-29 (Estimated); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All patients will also have blood samples drawn for genetic analysis and potential biomarker testing at Day 0 or at another visit during the study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Open Angle Glaucoma: • Group A (diagnosis of primary open-angle glaucoma or pseudo-exfoliative glaucoma) - subjects with documented disease progression in the past and high IOP (IOP above target), disc hemorrhage, family history of glaucoma-related vision loss or thin central cornea (<510um),
  * Progression is confirmed with repeatable abnormal standard automated perimetry (SAP) or progressive glaucomatous optic neuropathy
  * For patients that have had previous glaucoma surgery, they can be included if they have had documented glaucomatous progression post-surgery
  * Best corrected visual acuity of 20/40 or better at enrollment
- Healthy Individuals: • Group B (healthy controls)- healthy subjects without any ophthalmic disease and an IOP < 22mmHg
  o Normal appearing optic disc and no evidence of optic disc damage

SUMMARY:
The purpose of this study is to perform exploratory analyses to evaluate rates of functional and structural change in glaucoma, to identify predictors of rapid progression in patients with glaucoma and to identify possible genetic factors and biomarkers associated with the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

To identify and combine a set of predictors (i.e. by statistical modeling, machine learning classifiers or neural networks) to predict progression in glaucoma patients To determine how to most sensitively and specifically determine progression for a trial of a potential neuroprotective agent.

SECONDARY OBJECTIVES

To evaluate genetic and other potential biomarkers associated with progression in glaucoma.

To evaluate tests currently used on glaucoma patients to better predict which ones are most sensitive to detect disease progression and measure rates of change.

To assess progression by structural and functional tests:

* Optic disc stereophotographs
* Cirrus OCT
* RTVue OCT
* Standard Automated Perimetry (SAP)
* Frequency Doubling Technology Matrix

ELIGIBILITY:
INCLUSION CRITERIA

Subjects will be eligible if the following criteria are met:

* Group A (diagnosis of primary open-angle glaucoma or pseudo-exfoliative glaucoma) - subjects with documented disease progression in the past 3 years and high IOP (IOP above target), disc hemorrhage (within 3 years), family history of glaucoma-related vision loss or thin central cornea (<510um),

  * Progression is confirmed with repeatable abnormal standard automated perimetry (SAP) or progressive glaucomatous optic neuropathy
  * For patients that have had previous glaucoma surgery, they can be included if they have had documented glaucomatous progression post-surgery
  * Best corrected visual acuity of 20/40 or better at enrollment
* Group B (healthy controls)- healthy subjects without any ophthalmic disease and an IOP < 22mmHg

  o Normal appearing optic disc and no evidence of optic disc damage
* Ability to provide written informed consent for participation in this study

EXCLUSION CRITERIA

Subjects who meet any of the following criteria will be excluded from this study:

* Subjects with an ocular disease other than glaucoma
* Subjects participating in a long-term interventional clinical trial
* Subjects with any other medical condition which would prohibit them from making all study visits within the 24 months
* Glaucoma patients who have not demonstrated disease progression in the past 3 years
* Patients with diagnosis of pigmentary dispersion syndrome/glaucoma
* Patients that have had glaucoma surgery and have IOP ≤ 12 mm Hg
* Patients with advanced glaucoma with MD ≤ -20 dB
* Patients with a history of LASIK surgery
* Patients with myopia > -6.0 diopters.
* Patients with hyperopia >+6.0 diopters.
* In the investigator's opinion, any patient that cannot satisfactorily complete all of the structural and functional testing included in the protocol (investigator determined)
* Unable to perform reliable VF testing (Fixation losses 33% or less, false negative rate 33% or less and false positive rate of 15% or less) at the time of study entry
* In the investigator's opinion, any patient with an ocular disease that could impact study assessments
* Patients with cataracts in which surgery is planned or anticipated within the next 3 months.
* Patients with narrow angles in which laser iridotomy is planned or anticipated within the next 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Open Angle Glaucoma Health Individuals
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Weinreb, MD, Principal Investigator — UCSD Shiley Eye Institute
Locations (1):
- Hamilton Glaucoma Center, UCSD, La Jolla, California, United States

REFERENCES:
- [Background] Medeiros FA, Alencar LM, Zangwill LM, Sample PA, Weinreb RN. The Relationship between intraocular pressure and progressive retinal nerve fiber layer loss in glaucoma. Ophthalmology. 2009 Jun;116(6):1125-33.e1-3. doi: 10.1016/j.ophtha.2008.12.062. Epub 2009 Apr 19. PMID 19376584
- [Background] Medeiros FA, Alencar LM, Sample PA, Zangwill LM, Susanna R Jr, Weinreb RN. The relationship between intraocular pressure reduction and rates of progressive visual field loss in eyes with optic disc hemorrhage. Ophthalmology. 2010 Nov;117(11):2061-6. doi: 10.1016/j.ophtha.2010.02.015. Epub 2010 Jun 11. PMID 20541265
- [Background] Medeiros FA, Zangwill LM, Alencar LM, Bowd C, Sample PA, Susanna R Jr, Weinreb RN. Detection of glaucoma progression with stratus OCT retinal nerve fiber layer, optic nerve head, and macular thickness measurements. Invest Ophthalmol Vis Sci. 2009 Dec;50(12):5741-8. doi: 10.1167/iovs.09-3715. Epub 2009 Oct 8. PMID 19815731
- [Background] Alencar LM, Zangwill LM, Weinreb RN, Bowd C, Vizzeri G, Sample PA, Susanna R Jr, Medeiros FA. Agreement for detecting glaucoma progression with the GDx guided progression analysis, automated perimetry, and optic disc photography. Ophthalmology. 2010 Mar;117(3):462-70. doi: 10.1016/j.ophtha.2009.08.012. Epub 2009 Dec 24. PMID 20036010